CLINICAL TRIAL: NCT04856384
Title: Understanding the Effect of Variances on Precision in Predictive Coding When Walking to Music and Metronomes in Persons With Multiple Sclerosis With Progressive Subtypes.
Brief Title: Effect of Variance on Error Correction During Coupling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: National MS Center Melsbroek (Other); Revalidatie & MS Centrum Overpelt (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MS-Music-LM-001
Record Dates: First submitted 2021-01-29; First posted 2021-04-23 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis; Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- persons with Multiple Sclerosis (Experimental)
  Interventions: Other: synchronisation abilities
- Healthy controls (Experimental)
  Interventions: Other: synchronisation abilities

INTERVENTIONS:
Other: synchronisation abilities — The study contains 1 descriptive and 3 experimental sessions. In the descriptive session, participant's clinical motor and cognitive functions are collected. In the first experimental session, participant's beat perception and synchronisation abilities is examined within a finger tapping paradigm. In the following experimental sessions participants synchronsiation abilities is examined during walking paradigms, to music and metronomes, with period and phase auditory manipulations

SUMMARY:
This study is a case-control study, involving persons with progressive multiple sclerosis and healthy controls. The study contains 1 descriptive and 3 experimental sessions. In the descriptive session, participant's clinical motor and cognitive functions are collected. In the first experimental session, participant's beat perception and synchronisation abilities is examined within a finger tapping paradigm. In the following experimental sessions participants synchronsiation abilities is examined during walking paradigms, to music and metronomes, with period and phase auditory manipulations. In the latter twp sessions, apart from outcome measures of synchronization the following will be collected as well: brain activity using EEG recordings, spatio-temporal gait parameters, perceived fatigue, perceived motivation and perceived speed of walking.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Multiple sclerosis >1 year, diagnosis of progressive MS,
* walking speed 0.8-1.2m/s, ability to walk for 6 minutes continuously (canes and rollators are permitted)

Exclusion Criteria:

* relapse 3 months prior to enrollment,
* cognitive impairment impeding understanding of instructions,
* beat amusia,
* deafness,
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Motricity Index of dorsi flexors, knee extensors and hip flexors | baseline
  Muscle weakness
Modified Aschowrth scale Hamstrings, Tricepts Surae, Quadricepts | baseline
  Spasticity
Scale for the assessment and rating of ataxia | Baseline
  ataxia
Dynamic gait index | Baseline
  dynamic balance
Time up and Go test | Baseline
  Balance
6 minute walking test | Baseline
  gait pattern and endurance
Brief repeatable battery of Rao | Baseline
  cognitive test
Symbol digit mobility test | Baseline
  cognitive test
Stroop test 0 | Baseline
  cognitive test
MS walking scale -12 | Baseline
  impact of MS on walking ability
Activities-specific balance confidence scale | Baseline
  rating of balance confidence in performing activities of daily life
Modified fatigue impact scale | baseline
  effect of fatigue
Hospital Anxiety and Depression Scale | Baseline
  determine the levels of anxiety and depression
Dual task questionnaire | Baseline
  troubles a person have when performing a dual task during daily activity
Perceptual tempo and rhythm judgements | week 1
  subjective indications in regards to what the participants hear in terms
Asynchrony | week 1
  timing difference between the tap and the beat
64 channel EEG measurement | week 1
  neural correlates of entrainment
Resultant Vector Length | week 2
  synchronisation consistency
Resultant Vector Length | week 3
  synchronisation consistency
Relative phase angle | week 2
  asynchrony in time to quantify synchronization accuracy (in degrees and in milliseconds respectively)
Relative phase angle | week 3
  asynchrony in time to quantify synchronization accuracy (in degrees and in milliseconds respectively)

SECONDARY OUTCOMES:
Cadencce | week 2
  number of steps per minute
Cadencce | week 3
  number of steps per minute
Stride length | week 2
  distance between consecutive steps (cm)
Stride length | week 3
  distance between consecutive steps (cm)
Speed | week 2
  gait velocity (m/s)
Speed | week 3
  gait velocity (m/s)
Double Support | week 2
  time that both legs are in contact with the floor (mseconds)
Double Support | week 3
  time that both legs are in contact with the floor (mseconds)
Perceived cognitive and physical fatigue | week 2
  A visual analogue scale will be used, and participants will be asked to rate their perceived cognitive and physical fatigue levels before and after each experimental walking conditions
Perceived cognitive and physical fatigue | week 3
  A visual analogue scale will be used, and participants will be asked to rate their perceived cognitive and physical fatigue levels before and after each experimental walking conditions
Perceived motivation | week 2
  A Likert scale will be used, and participants will be asked to rate their perceived motivation of walking after each experimental walking conditions
Perceived motivation | week 3
  A Likert scale will be used, and participants will be asked to rate their perceived motivation of walking after each experimental walking conditions
Perceived walking speed | week 2
  A Likert scale will be used, and participants will be asked to rate their perceived walking speed relative to their usual walking after each experimental walking conditions
Perceived walking speed | week 3
  A Likert scale will be used, and participants will be asked to rate their perceived walking speed relative to their usual walking after each experimental walking conditions
64 channel EEG measurement (only conducted in 4 PwMS and HC) | week 2
  Neural correlates of entrainment
64 channel EEG measurement (only conducted in 4 PwMS and HC) | week 3
  Neural correlates of entrainment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, prof. dr., Principal Investigator — Hasselt University; Lousin Moumdjian, dr., Study Chair — Hasselt University
Locations (2):
- Belgium (2):
  - National MS Center Melsbroek, Melsbroek
  - Noorderhart Revalidatie & MS centrum, Overpelt

IPD SHARING:
Plan to Share IPD: No